CLINICAL TRIAL: NCT01205269
Title: A Double-blind, Placebo-controlled, Randomised, Multi-centre, 3-way Cross-over, Single-dose Phase II Study to Investigate the Local and Systemic Effects of Inhaled AZD8683 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: The Study Will Evaluate the Effect of AZD8683 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D1883C00004; EudraCT number: 2010-020506-15
Record Dates: First submitted 2010-09-15; First posted 2010-09-20 (Estimated); Results first posted 2013-11-13 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease (COPD); safety; inhalation; long-acting muscarinic receptor antagonist (LAMA)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- First 50 mcg, then 200 mcg, then placebo (Experimental): period 1: AZD8683 50 mcg, period 2: washout, period 3: AZD8683 200 mcg, period 4:washout, period5: placebo
  Interventions: Drug: AZD8683, 50 mcg; Drug: Placebo; Drug: AZD8683, 200 mcg
- First 50 mcg, then placebo, then 200 mcg (Experimental): period 1: AZD8683 50 mcg, period 2: washout, period 3: placebo, period 4: washout, period5:AZD8683 200 mcg
  Interventions: Drug: AZD8683, 50 mcg; Drug: Placebo; Drug: AZD8683, 200 mcg
- First 200 mcg, then placebo, then 50 mcg (Experimental): period 1: AZD8683 200 mcg, period 2: washout, period 3: placebo, period 4: washout, period 5: AZD8683 50 mcg
  Interventions: Drug: AZD8683, 50 mcg; Drug: Placebo; Drug: AZD8683, 200 mcg
- First 200 mcg, then 50 mcg, then placebo (Experimental): period 1: AZD8683 200 mcg, period 2: washout, period 3: AZD8683 50 mcg, period 4: washout, period 5: placebo
  Interventions: Drug: AZD8683, 50 mcg; Drug: Placebo; Drug: AZD8683, 200 mcg
- First placebo, then 200 mcg, then 50 mcg (Experimental): period 1: placebo , period 2: washout, period 3: AZD8683 200 mcg, period 4: washout, period5: AZD8683 50 mcg
  Interventions: Drug: AZD8683, 50 mcg; Drug: Placebo; Drug: AZD8683, 200 mcg
- First placebo, then 50 mcg, then 200 mcg (Experimental): period 1: placebo , period 2: washout, period 3: AZD8683 50 mcg, period 4: washout, period5: AZD8683 200 mcg
  Interventions: Drug: AZD8683, 50 mcg; Drug: Placebo; Drug: AZD8683, 200 mcg

INTERVENTIONS:
Drug: AZD8683, 50 mcg — Dry powder for inhalation, single dose
Drug: Placebo — Dry powder for inhalation, single dose
Drug: AZD8683, 200 mcg — Dry powder for inhalation, single dose

SUMMARY:
The purpose of this study is to investigate effects of inhaled AZD8683 compared to placebo in COPD patients.

DETAILED DESCRIPTION:
A double-blind, placebo-controlled, randomised, multi-centre, 3-way cross-over, single-dose phase II study to investigate the local and systemic effects of inhaled AZD8683 in patients with chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD
* Current or ex-smokers
* FEV1 40 - 80% of the predicted normal value (post-bronchodilator) and post-bronchodilator FEV1/FVC < 70%

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically relevant abnormal findings at screening examinations
* Family history or presence of glaucoma
* Need of long term oxygen therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kuna, MD Professor, Principal Investigator — Poland
Locations (4):
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Lodz
  - Research Site, Proszowice

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study has been performed at four centers in Poland. The first subject entered the study on 10 October 2010 and the last subject completed the study on 17 December 2010. The randomised population consisted of 28 patients, 27 completed the study. All patients were included in the analysis of all variables.
Groups:
- First 50 mcg, Then 200 mcg, Then Placebo: period 1: AZD8683 50 mcg, period 2: washout, period 3: AZD8683 200 mcg, period 4: washout, period5: placebo
Period: Period 1 - First Intervention
Arm/Group | First 50 mcg, Then 200 mcg, Then Placebo | First 50 mcg, Then Placebo, Then 200 mcg | First 200 mcg, Then Placebo, Then 50 mcg | First 200 mcg, Then 50 mcg, Then Placebo | First Placebo, Then 200 mcg, Then 50 mcg | First Placebo, Then 50 mcg, Then 200 mcg
Started | 4 | 4 | 4 | 6 | 5 | 5
Completed | 4 | 4 | 4 | 6 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 - Washout
Arm/Group | First 50 mcg, Then 200 mcg, Then Placebo | First 50 mcg, Then Placebo, Then 200 mcg | First 200 mcg, Then Placebo, Then 50 mcg | First 200 mcg, Then 50 mcg, Then Placebo | First Placebo, Then 200 mcg, Then 50 mcg | First Placebo, Then 50 mcg, Then 200 mcg
Started | 4 | 4 | 4 | 6 | 5 | 5
Completed | 4 | 4 | 4 | 6 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 - Second Intervention
Arm/Group | First 50 mcg, Then 200 mcg, Then Placebo | First 50 mcg, Then Placebo, Then 200 mcg | First 200 mcg, Then Placebo, Then 50 mcg | First 200 mcg, Then 50 mcg, Then Placebo | First Placebo, Then 200 mcg, Then 50 mcg | First Placebo, Then 50 mcg, Then 200 mcg
Started | 4 | 4 | 4 | 6 | 5 | 5
Completed | 4 | 4 | 4 | 6 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 - Washout
Arm/Group | First 50 mcg, Then 200 mcg, Then Placebo | First 50 mcg, Then Placebo, Then 200 mcg | First 200 mcg, Then Placebo, Then 50 mcg | First 200 mcg, Then 50 mcg, Then Placebo | First Placebo, Then 200 mcg, Then 50 mcg | First Placebo, Then 50 mcg, Then 200 mcg
Started | 4 | 4 | 4 | 6 | 5 | 5
Completed | 4 | 4 | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Eligibility criteria not fulfilled | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 5 - Third Intervention
Arm/Group | First 50 mcg, Then 200 mcg, Then Placebo | First 50 mcg, Then Placebo, Then 200 mcg | First 200 mcg, Then Placebo, Then 50 mcg | First 200 mcg, Then 50 mcg, Then Placebo | First Placebo, Then 200 mcg, Then 50 mcg | First Placebo, Then 50 mcg, Then 200 mcg
Started | 4 | 4 | 4 | 5 | 5 | 5
Completed | 4 | 4 | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all groups randomized to one of 6 sequences of drug or placebo.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 28
Age, Continuous [Mean (Full Range); unit: years] | 63.2 [52 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1), Peak Effect Within 0 - 24 Hours Post-dose
Description: Maximum FEV1 value
Time Frame: 0, 5 min, 15 min, 30 min, 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, 12 h, 14 h, 18 h, 22 h, 24 h
Population: Of the 28 randomised patients, 27 completed the study and one discontinued during the last washout period. All 28 randomised patients were included in the analyses of all variables
Measure: Mean (Standard Deviation); unit: L
Groups:
- AZD8683 50 mcg: 1 x AZD8683 Turbuhaler 50mcg + 3x placebo Turbuhaler (dry powder inhaler)
- AZD8683 200 mcg: 1 x AZD8683 Turbuhaler 50 mcg + 3 x AZD8683 Turbuhaler 50 mcg (dry powder inhaler)
- Placebo: 1 x Placebo Turbuhaler + 3 x Placebo Turbuhaler (dry powder inhaler)
Arm/Group | AZD8683 50 mcg | AZD8683 200 mcg | Placebo
Number analyzed (Participants) | 28 | 28 | 27
L | 1.67 (0.48) | 1.73 (0.47) | 1.64 (0.47)

2. Primary Outcome: Forced Expiratory Volume in One Second (FEV1), Average Effect Over 22 - 26 Hours Post-dose
Description: Trough FEV1 value
Time Frame: 22 h, 24 h, 26 h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD8683 50 mcg | AZD8683 200 mcg | Placebo
Number analyzed (Participants) | 28 | 28 | 27
L | 1.53 (0.46) | 1.60 (0.46) | 1.49 (0.46)

3. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1), Average Effect Over 0 - 24 Hours Post-dose
Description: Average FEV1 value
Time Frame: 0, 5 min, 15 min, 30 min, 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, 12 h, 14 h, 18 h, 22 h, 24 h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD8683 50 mcg | AZD8683 200 mcg | Placebo
Number analyzed (Participants) | 28 | 28 | 27
L | 1.49 (0.42) | 1.54 (0.42) | 1.44 (0.42)

4. Secondary Outcome: Forced Vital Capacity (FVC), Peak Effect Over 0 - 24 Hours Post-dose
Description: Maximum FVC value
Time Frame: 0, 5 min, 15 min, 30 min, 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, 12 h, 14 h, 18 h, 22 h, 24 h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD8683 50 mcg | AZD8683 200 mcg | Placebo
Number analyzed (Participants) | 28 | 28 | 27
L | 3.35 (0.87) | 3.39 (0.81) | 3.28 (0.78)

5. Secondary Outcome: Systolic Blood Pressure, Average Effect Over 0 - 4 Hours Post-dose
Description: Average systolic blood pressure value
Time Frame: 0, 30 min, 2 h, 4 h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD8683 50 mcg | AZD8683 200 mcg | Placebo
Number analyzed (Participants) | 28 | 28 | 27
mmHg | 130.7 (14.1) | 131.2 (12.0) | 132.2 (13.3)

6. Secondary Outcome: Diastolic Blood Pressure, Average Effect Over 0 - 4 Hours Post-dose
Description: Average diastolic blood pressure value
Time Frame: 0, 30 min, 2 h, 4 h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD8683 50 mcg | AZD8683 200 mcg | Placebo
Number analyzed (Participants) | 28 | 28 | 27
mmHg | 77.9 (7.6) | 77.5 (6.5) | 77.7 (7.9)

7. Secondary Outcome: Pulse, Average Effect Over 0 - 4 Hours Post-dose
Description: Average pulse value
Time Frame: 0, 30 min, 2 h, 4 h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | AZD8683 50 mcg | AZD8683 200 mcg | Placebo
Number analyzed (Participants) | 28 | 28 | 27
bpm | 77.3 (10.5) | 76.0 (11.9) | 74.9 (9.5)

8. Secondary Outcome: Heart Rate, Average Effect Over 0 - 4 Hours Post-dose
Description: Average heart rate value
Time Frame: 0, 30 min, 2 h, 4 h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | AZD8683 50 mcg | AZD8683 200 mcg | Placebo
Number analyzed (Participants) | 28 | 28 | 27
bpm | 76.2 (12.1) | 75.0 (13.4) | 72.8 (11.4)

9. Secondary Outcome: QTcF, Average Effect Over 0 - 4 Hours Post-dose
Description: Average QTcF value. QTcF = QT interval corrected for heart rate using Fridericia's formula
Time Frame: 0, 30 min, 2 h, 4 h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | AZD8683 50 mcg | AZD8683 200 mcg | Placebo
Number analyzed (Participants) | 28 | 28 | 27
ms | 412.8 (22.4) | 409.1 (23.7) | 411.9 (22.0)

10. Secondary Outcome: Plasma AZD8683 Cmax
Description: Maximum plasma concentration of AZD8683
Time Frame: 0, 5 min, 15 min, 30 min, 45 min, 1 h, 90 min, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h
Population: Plasma concentrations were below the LLOQ for all post-dose samples for some patients and treatments. PK parameters for these 3 treatments have been set to missing and are not included in the descriptive statistics.
Measure: Geometric Mean (Full Range); unit: nmol/L
Arm/Group | AZD8683 50 mcg | AZD8683 200 mcg | Placebo
Number analyzed (Participants) | 26 | 27 | 0
nmol/L | 0.0578 [0.008 to 0.262] | 0.2791 [0.030 to 1.250] |

11. Secondary Outcome: Plasma AZD8683 AUC0-24
Description: Area under the AZD8683 plasma concentration curve from 0 to 24 hours
Time Frame: 0, 5 min, 15 min, 30 min, 45 min, 1 h, 90 min, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: nmol*h/L
Arm/Group | AZD8683 50 mcg | AZD8683 200 mcg | Placebo
Number analyzed (Participants) | 26 | 27 | 0
nmol*h/L | 0.1872 [0.013 to 0.836] | 0.8427 [0.104 to 2.764] |

ADVERSE EVENTS:
Arm/Group | AZD8683 50 mcg | AZD8683 200 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AZ for review at least 60 days in advance of submission for publication. Investigators in multicenter (MC) studies agree to postpone MC publications until the earlier of the date of the first AZ-authorized MC publication or a period up to 18 months from study completion at all sites. AZ has the right to request delays: up to 60 days for confidential information, and an additional 90 days to protect intellectual property.